CLINICAL TRIAL: NCT04082728
Title: Evaluation of the Added Value of Metamizole to Standard Post-operative Treatment After Ambulant Surgery: a Double-blind, Randomized, Controlled Trial
Brief Title: Evaluation of the Added Value of Metamizole to Standard Post-operative Treatment After Ambulant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Anesthesiologist, MD, PhD, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Metamizole002
Record Dates: First submitted 2019-09-02; First posted 2019-09-09 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Analgesia; Surgery; Recovery
Keywords: ambulant surgery; post-operative medication; recovery
MeSH Terms: conditions — Agnosia | interventions — Dipyrone

STUDY DESIGN:
Intervention Model Description: This trial is designed as a mono-center, prospective, double-blind, randomized placebo controlled superiority trial comparing 2 groups of patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metamizole (Active Comparator): Patients in the experimental group will be instructed to take metamizole 1000 mg orally three times a day for four days, ibuprofen 600 mg orally three times a day for four days and 1000 mg paracetamol orally four times a day during the entire study period.
  Interventions: Drug: Metamizole
- Placebo (Placebo Comparator): Patients in the experimental group will be instructed to take a placebo orally three times a day for four days, ibuprofen 600 mg orally three times a day for four days and 1000 mg paracetamol orally four times a day during the entire study period.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Metamizole — Patients in the experimental group will be instructed to take metamizole 1000 mg orally three times a day for four days. All patients will be instructed to take ibuprofen 600 mg orally three times a day for four days and 1000 mg paracetamol orally four times a day during the entire study period.
  Arms: Metamizole
Drug: Placebo oral tablet — Patients in the placebo group will be instructed to take a placebo orally three times a day for four days. All patients will be instructed to take ibuprofen 600 mg orally three times a day for four days and 1000 mg paracetamol orally four times a day during the entire study period.
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate if the addition of metamizole to the standard post-operative treatment, i.e. paracetamol and ibuprofen, is superior in reducing post-operative pain on day 1 after ambulatory surgery compared to the standard post-operative treatment.

Therefore, a mono-center, prospective, double-blind, randomized controlled superiority trail will be designed in order to investigate superiority of metamizole compared to the standard post-operative treatment in patients undergoing arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
Ambulant surgery has been expanding substantially in the past decade, primarily because it is associated with lower costs and it is believed to be as safe as surgery in the in-patient setting. Moreover, it seems that early discharge can contribute to a faster recovery and a decreased incidence of hospital-associated complications. In view of the relative absence of major complications, post-operative pain and quality of recovery should be considered the principal endpoints after day surgery. The quality of recovery after different types of surgery is of major importance since the evaluation of recovery allows a discrimination between a normal and pathological health trajectory. A disadvantage in the ambulatory setting is related to the absence of postoperative surveillance by professionals. This implicates that the individual patient has to assess, without any support, if his/her quality of recovery is normal or not. There is limited information on procedure-specific quality of recovery after day surgery, however, different tools such as the 1-tem Global Surgical Recovery (GSR) index and the 5-dimensional European Quality of Life (EQ5D) questionnaires can be addressed.

Particularly in the ambulant setting, good post-operative analgesia is challenging because patients have to control pain at home by themselves, in the absence of hospital staff. Moreover, there is a limit in the type of analgesia that is available (i.e. no strong opioids) as well as in the route of administration (i.e. no epidural, intravenous, subcutaneous or intramuscular route) at home. Nowadays a multimodal approach to control pain has been advocated in the ambulatory setting. This approach is based on a combination of paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs) and, if necessary, weak opioids. A local and regional anesthesia also have been advocated in the ambulatory setting to relieve pain for 8 to 24 hours after surgery. Despite this multimodal pain therapy, the prevalence of outpatients suffering moderate to severe acute postoperative pain at home still remains high and varies from 9 to 40%. More specific, patients undergoing haemorrhoid surgery, arthroscopic shoulder and knee surgery, and inguinal hernia repair seem to be at highest risk to develop moderate to severe pain on the fourth postoperative day.

Due to this relatively high prevalence and due to the fact that NSAIDs are not always sufficiently effective, can have numerous contraindications and therefore are not suitable in up to 25% of all patients; there is a need for an alternative pain therapy.

Metamizole (dipyrone) is a non-opioid compound with strong analgesic, antipyretic and spasmolytic effects. The analgesic efficacy of intravenous or intramuscular metamizole for pain relief after inpatient surgery is well described. Recently, we showed in a prospective, double-blind, randomized controlled trial that the combination of paracetamol and metamizole is equally effective in treatment of acute post-operative pain at home after ambulatory surgery compared to paracetamol and ibuprofen. Moreover, patient satisfaction was equal in both groups, as well as the reported side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years
* ASA classification 1,2 or 3
* Body weight > 50 kg
* Undergoing ambulatory arthroscopic shoulder surgery (SAD ± ACJ excision or decompression, decompression + biceps tenodesis, rotator cuff repair, rotator cuff repair + decompression (+ biceps tenodesis)

Exclusion Criteria:

* Not meeting inclusion criteria
* Patients undergoing SLAP of Bankart repair
* Cognitive impairment or no understanding of the Dutch language
* Preoperative pharmacological pain treatment and/or a history of chronic pain
* Allergy to or contraindication for taking the study medication (e.g. paracetamol, metamizole, ibuprofen or another non-steroidal anti-inflammatory drug)
* Porphyria
* Pregnancy or lactation
* A history of severe renal, hepatic, pulmonary or cardiac failure
* Current symptoms or a history of gastrointestinal bleeding
* Ileus or chronic obstipation
* A history of substance abuse, or use of medication with a suppressive effect on the central nervous system
* Hypotension
* Hematological disease
* Use of anti-rheumatic drugs
* Rhinosinusitis or nasal polyposis
* Glucose-6-phosphate dehydrogenase deficiency
* Fever or other signs of infection
* Refusal of an interscalene block

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Postoperative pain on day 1 | 24 hours after the surgery
  Postoperative pain intensity at movement measured by an 11-point Numeric Rating Scale (NRS) where 0: no pain and 10: worst imaginary pain) on postoperative day 1.

SECONDARY OUTCOMES:
Quality of recovery | at baseline and days 7, 14, 28 and 3 months postoperatively.
  Quality of Recovery measured by the 1-item Global Surgical Recovery (GSR) index which represents a single question about the extent to which patients consider themselves to be recovered from surgery (0-100%) at baseline and days 7, 14, 28 and 3 months postoperatively.
Quality of recovery | at baseline and days 7, 14, 28 and 3 months postoperatively.
  Measured with the EuroQol (EQ5D) questionnaire, which is non-disease specific instrument developed for describing and valuing health-related quality of life, at baseline and days 7, 14, 28 and 3 months postoperatively.
Postoperative pain | at baseline, at discharge and at day 1, 2, 3, 4, 7, 14, 28 and at 3 months after surgery
  Postoperative pain intensity at rest and at movement measured by an 11-point Numeric Rating Scale (NRS) where 0: no pain and 10: worst imaginary pain) at baseline, at discharge and at day 1, 2, 3, 4, 7, 14, 28 and at 3 months.
Simple Shoulder test | at baseline and days 7, 14, 28 and 3 months postoperatively.
  Simple shoulder test (SST) measured at baseline and days 7, 14, 28 and 3 months postoperatively.
Adherence | day 1, 2, 3 and 4 postoperatively.
  Adherence to study medication on day 1, 2, 3 and 4 postoperatively. Definition compliance: Full compliance: analgesia used as prescribed "yes", no compliance: analgesia used as prescribed "no"
Piritramide | after surgery until discharge of PACU (up to 3 hours after surgery)
  Total amount of intravenous piritramide received in the post-operative care unit (PACU)
Rescue medication | day 1, 2, 3 and 4 postoperatively
  The use of rescue medication (Tramadol) at home on day 1, 2, 3 and 4 postoperatively (yes/no)
Satisfaction with study medication, surgery and hospital care and telephone follow-up | at day 7 and 3 months postoperative
  Satisfaction with study medication, surgery and hospital care and telephone follow-up measured at day 7 and 3 months postoperative measured by an 11-point Numeric Rating Scale (NRS) where 0: totally unsatisfied and 10: totally satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stessel B, Lambrechts M, Evers S, Vanderstappen C, Callebaut I, Ory JP, Herbots J, Dreesen I, Vaninbroukx M, Van de Velde M. Additive or synergistic analgesic effect of metamizole on standard pain treatment at home after arthroscopic shoulder surgery: A randomised controlled superiority trial. Eur J Anaesthesiol. 2023 Mar 1;40(3):171-178. doi: 10.1097/EJA.0000000000001792. Epub 2023 Jan 11. PMID 36632758